CLINICAL TRIAL: NCT06105645
Title: Contribution of Fast-ripples to the Improvement of the Neurosurgical Management of Drug-refractory Epilepsy
Acronym: NENUFAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Centre de recherche Cerveau et Cognition (CERCO) (Unknown); Dixi Medical (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC31/22/0260; 2022-A02552-41 (Other: ID-RCB)
Record Dates: First submitted 2023-10-23; First posted 2023-10-27 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Epilepsy
Keywords: Fast-ripples; Epilepsy; Neurosurgery; Hybrid electrodes; MICRODEEP® MME hybrid electrodes; StereoEEG
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm with fast-ripples information (Experimental): Patients for whom 4-6 usual clinical macro-electrodes will be replaced by hybrid micro-macro electrodes and for whom fast-ripples will be assessed
  Interventions: Device: DIXI Medical Microdeep® Micro- Macro Depth electrodes
- Arm without fast-ripples information (Active Comparator): Patients who will undergo an SEEG with the usual electrodes and for whom fast-ripples will not be assessed.
  Interventions: Device: Standard electrodes

INTERVENTIONS:
Device: DIXI Medical Microdeep® Micro- Macro Depth electrodes — It is a deep intracerebral electrode used in the pre-surgical diagnosis of certain drug-resistant epilepsies. It consists of micro- and macro-contacts and is designed for Stereo-ElectroEncephalography (SEEG) recording via the macro-contacts or micro-contacts and brief stimulation via the macro-contacts.
  Arms: Arm with fast-ripples information
Device: Standard electrodes — Standard electrodes used usually during the SEEG
  Arms: Arm without fast-ripples information

SUMMARY:
The main aim of this study is to evaluate the contribution of fast-ripples (FR) information on the neurosurgery management of patients with drug-refractory epilepsy investigated by Stereo-ElectroEncephaloGraphy (SEEG), as measured by freedom from disabling seizures one-year post-surgery.

220 patients (for whom 4-6 usual clinical macro-electrodes will be replaced by hybrid micro-macro electrodes and for whom fast-ripples will be assessed) distributed over 5 centres and 220 control patients(who will undergo an SEEG with the usual electrodes and for whom fast-ripples will not be assessed) distributed over 6 centres. This is a controlled, non-randomized, parallel plan, prospective, multicentre exploratory study.

DETAILED DESCRIPTION:
This is a controlled, non-randomized, parallel plan, prospective, multicentre exploratory study. The design of the study relies on two groups of patients benefiting from a SEEG, equivalent in size: one with standard and hybrid electrodes for which fast-ripple information will be available for the neurosurgery decision, the other, who will serve as a control group, with standard electrodes only and for which no information regarding fast-ripples will be provided. For all patients undergoing SEEG, the decisions about eligibility to epilepsy surgery and, if eligible, about the best surgical plan, are taken during a multidisciplinary epilepsy meeting (MEM) within the 4 +/- 2 months following the SEEG. In the group of patients with standard and hybrid electrodes, the procedure as extensively tested previously, is to plan the implantation of the standard electrodes as usually done, and once done, to replace from 4 to 6 standard electrodes with hybrid electrodes. In this group, intracerebral ElectroEncephaloGraphy (EEG) data will be acquired for detection of fast-ripples, during one hour of a rest period for 2 days during the first week of SEEG, as well as during one cycle of night sleep when possible. Fast-ripples(number, localization and characteristics) for all these patients will be analysed by an expert group of neuroscientists based in Toulouse blind to the analysis of the Epileptogenic Zone (EZ), irritative and propagation zones and on all micro- and macro contacts, to the participating centre and to the period of recording. The results of the fast-ripple assessment will be provided to the clinicians on time for the MEM. They will incorporate this information along other usual clinical information gathered during the SEEG to reach a conclusion regarding the possibility of a neurosurgery. No analysis of the fast-ripples will be performed in the other group of patients with standard electrodes only. In this group, the conclusion regarding the possibility of a neurosurgery will thus be done during the MEM with the standard clinical information gathered during the SEEG only. Following epilepsy surgery, the typical follow-up performed in routine in all participating centres includes a clinical evaluation one year after surgery, during which Engel class is assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patient suffering from drug-resistant focal epilepsy (DRFE), as defined by the International League Against Epilepsy, undergoing SEEG, the indication of which was selected during a multidisciplinary epilepsy meeting
* Patient who has given written informed consent to allow the study data collection procedures
* Patient covered by the French healthcare system.

Exclusion Criteria:

* Patients under juridical protection (authorship, curators or safeguarding of justice).
* Patient deprived of liberty by a judicial or administrative decision
* Patient with a cardiac defibrillator
* Thermocoagulation planned on one of the potential hybrid electrodes .
* Patient in exclusion period of another study.
* No other non-inclusion criteria since the study will only be proposed to patients who already meet the criteria for a SEEG

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2024-01-19 (Actual); Primary Completion 2030-04 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Contribution of fast-ripples information on freedom seizures | 12 months after epilepsy surgery
  Proportion of patients with Engel class I after one-year post-surgery in the group of patients with information of fast-ripples compared to patients without.

SECONDARY OUTCOMES:
Contribution of fast-ripples information on improvement of epilepsy | 12 months after epilepsy surgery
  Proportion of patients with Engel classes I to III one-year post-surgery of patients with information of fast-ripples compared to patients without.
Contribution of fast-ripples information on patients addressed to neurosurgery | 12 months after epilepsy surgery
  Proportion of patients operated for their epilepsy in the group of patients with information of fast-ripples compared to patients without.
Adverse effects related to Stereo-electroencephalography | Day 0 (SEEG visit)
  Quantitative and qualitative description of adverse effects related to the Stereo-electroencephalography (SEEG) in the group of patients with information of fast-ripples compared to patients without.
Adverse effects of epilepsy surgery | 6 months after surgical decision
  Quantitative and qualitative description of adverse effects related to epilepsy surgery in the group of patients with information of fast-ripples compared to patients without.
Adverse effects of hybrid electrodes | Day 0 (SEEG visit)
  Quantitative and qualitative description of adverse effects related to the hybrid electrodes.
Post-operative neurological deficit | 12 months after epilepsy surgery
  Number of patients suffering from disabling post-operative neurological deficit, anxiety or depression in the group of patients with information of fast-ripples versus patients without
Evolution of quality of life using the score of Quality of life Epilepsy Inventory Epilepsy Inventory | 12 months after epilepsy surgery
  Delta of quality of life using the score of Quality of life Epilepsy Inventory (QOLIE-31) between baseline and 12 months related to epilepsy surgery in the group of patients with information of fast-ripples compared to patients without.
  QOLIE-31 is a 31-item questionnaire with different proposal scores. The maximal total score is 100 : the higher the score, the better the quality of life
Level of satisfaction | 12 months after epilepsy surgery
  Mean of level of satisfaction with the outcome of epilepsy surgery assessed using the Evaluation of changes in daily life after epilepsy surgery (EVOCQUE) self-questionnaire, 12 months after surgery, related to epilepsy surgery in the group of patients with information of fast-ripples compared to patients without.
  EVOCQUE is a self-questionnaire with ten different questions and proposal scores.
Recording of fast-ripples | Day 0 (SEEG visit)
  Number of fast-ripples recorded on the hybrid electrodes, on the one hand on the micro- contacts and on the other hand on the adjacent macro-contacts of the same hybrid electrode.
Distribution of the fast-ripples | Day 0 (SEEG visit)
  Number of fast-ripples in the Epileptogenic Zone, Irritative Zone and healthy zone
Number of fast-ripples recorded according to the period | Day 0 (SEEG visit)
  Number of fast-ripples recorded during one period of sleep, an equivalent period of nap and an equivalent period of sitcom watching.

CONTACTS AND LOCATIONS:
Overall Officials: Luc VALTON, MD, Principal Investigator — University Hospital, Toulouse
Locations (11):
- France (11):
  - CHU Amiens Picardie, Amiens
  - University hospital of Bordeaux, Bordeaux
  - University hospital of Grenoble Alpes, La Tronche
  - APHP Hôpital Bicêtre, Le Kremlin-Bicêtre
  - CHU de Lille, Lille
  - Hospices Civils de Lyon, Lyon
  - CHRU de Nancy, Nancy
  - Fondation Adolphe de Rothschild, Paris
  - CHU de Rennes, Rennes
  - Hôpitaux universitaires de Strasbourg, Strasbourg
  - University Hospital of Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Despouy E, Curot J, Reddy L, Nowak LG, Deudon M, Sol JC, Lotterie JA, Denuelle M, Maziz A, Bergaud C, Thorpe SJ, Valton L, Barbeau EJ. Recording local field potential and neuronal activity with tetrodes in epileptic patients. J Neurosci Methods. 2020 Jul 15;341:108759. doi: 10.1016/j.jneumeth.2020.108759. Epub 2020 May 7. PMID 32389603